CLINICAL TRIAL: NCT05401851
Title: Bi-ventricular Epicardial Activation in Left Bundle Area Pacing: a Comparison Study
Acronym: LBBAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC-2022-020
Record Dates: First submitted 2022-04-04; First posted 2022-06-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-05

CONDITIONS: Bradyarrhythmia; Pacemaker Syndrome; Biventricular Cardiac Pacemaker Malfunction
Keywords: Left bundle area pacing; Pacemaker; Wide QRS
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Body surface mapping (Other): With the Insite Vest, activation of the epicardium will be performed.
  Interventions: Device: Left Bundel Area Pacing

INTERVENTIONS:
Device: Left Bundel Area Pacing — RV Lead will be placed deep in the interventricular septum

SUMMARY:
Study of the ventricular activation patterns during left bundle area pacing and compare it with baseline activation during normal sinus rhythm in patients with and without baseline bundle branch conduction disorder.

DETAILED DESCRIPTION:
Right ventricular (RV) pacing has long been the gold standard treatment for symptomatic brady arrhythmias. Right ventricular apical pacing has shown to cause electrical and mechanical desynchrony resulting in left ventricular (LV) dysfunction, and, in some cases, clinical heart failure together with other mechanical and arrhythmic complications. Hence, it was necessary to find a more physiologic method of pacing that ensures synchrony. His bundle pacing was first described in 2000, and is more recently adapted as a pacing method with less deleterious effects on the RV. However, lead dislodgement, high pacing thresholds, battery depletion, and difficulty identifying the exact location of His bundle were the most significant concerns related to this method. Subsequently, left bundle branch area pacing (LBB-AP), first described in 2017 by Huang et al, has emerged as safe alternative with excellent lead stability and capture threshold, and more ability to correct distal conduction disease as compared to His bundle pacing. Recent studies report promising mid-term outcome concerning left ventricular desynchrony. To the best of our knowledge, bi-ventricular activation was never studied in patients with LBB-AP.

Multiple tools have been used to assess biventricular (BiV) synchrony specially with chronic resynchronization therapy (CRT) including echocardiography and 12 lead ECG. Eschalier et al. found that epicardial noninvasive ECG mapping, was better at predicting clinical CRT response than QRS duration or the presence of LBBB. Activation patterns and timings with RV apical pacing, native LBBB, and BiV pacing have been well studied using this tool. With LBBP, however, these activation parameters have not yet been described.

This study aims to evaluate bi-ventricular activation in patients equipped with LBB-AP using non-invasive 3D mapping system in patients with or without baseline ventricular conduction disorder.

ELIGIBILITY:
Inclusion Criteria:

* 30 patients with a functional LBB-AP pacemaker

Exclusion Criteria:

* Age < 18 years
* Previous cardiac surgery
* Cardiomyopathy with documented ventricular scar
* Patients with prior pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-02-21 (Estimated); Study Completion 2024-10-21 (Estimated)

PRIMARY OUTCOMES:
Epicardial map | 1 day
  Activation patterns (visual inspection) on non-invasive 3D ECG mapping
Epicardial map | 1 day
  Activation time (ms) on non-invasive 3D ECG mapping

SECONDARY OUTCOMES:
Echo parameters for resynchronization | 90 days
  LVEF (%)
Echo parameters for resynchronization | 90 days
  intraventricular delay (ms)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo De Asmundis, MD, PhD, Principal Investigator — UZ Brussels
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No